CLINICAL TRIAL: NCT01583972
Title: Efficacy of Newborn Vitamin A Supplementation in Improving Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N3-TSA-003; PR-10012 (Other: icddr.b)
Record Dates: First submitted 2012-04-14; First posted 2012-04-24 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Vitamin A Deficiency
Keywords: Vitamin A deficiency; Vitamin A; retinyl palmitate; malnutrition; vaccine; vaccination; BCG; tuberculosis; polio virus; tetanus toxoid; hepatitis B virus; thymus; T lymphocyte; B lymphocyte; antibody; bacterial translocation; T-cell receptor excision circle
MeSH Terms: conditions — Vitamin A Deficiency; Malnutrition; Tuberculosis; Tetanus; Hepatitis B | interventions — retinol palmitate; Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin A (Experimental): 50,000 IU vitamin A in edible oil
  Interventions: Dietary Supplement: retinyl palmitate
- Placebo (Placebo Comparator): edible oil used as diluent for vitamin A
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: retinyl palmitate — 50,000 IU vitamin A in oil given within 48 h of birth from single-dose capsule
  Other Names: Vitamin A
  Arms: Vitamin A
Dietary Supplement: Placebo — edible oil used as diluent for vitamin A given within 48 h of birth from single-dose capsule identical in appearance to vitamin A capsule
  Arms: Placebo

SUMMARY:
Vitamin A supplementation at birth may increase survival of infants through one year of age by reducing mortality from infectious diseases, though current studies are not conclusive on this point. The goal of our study is to determine if supplementation of newborn infants with 50,000 IU of vitamin A improves aspects of immune function that may be impaired by vitamin A deficiency. Our underlying assumption is that supplementation may thus decrease risk of death by improving immune function and the ability to survive infections. This project will be limited to the examination of the impact of vitamin A on immune function and will not aim to determine the impact on morbidity or mortality, which would require larger sample sizes. The hypotheses addressed by this study are as follows: Provision of vitamin A supplements to newborns at risk of vitamin A deficiency will (1) improve functioning of the thymus (the source of T lymphocytes, cells of the immune system that are important in response to infection and immunization); (2) enhance T lymphocyte-mediated responses to standard vaccines given at birth and early in infancy; and (3) improve gut barrier function (i.e., ability to prevent bacterial infection across the epithelial barrier), relative to provision of a placebo.

DETAILED DESCRIPTION:
This project will examine the effect of vitamin A supplementation (50,000 IU) or placebo given with BCG and oral polio virus (OPV) immunization within 48 h of birth on immune function in 300 Bangladeshi infants (150 in each group) at risk of vitamin A deficiency recruited in a poor community of Dhaka, Bangladesh. Infants will be followed from birth through 15 wk of age. Current evidence from community-based mortality trials is not conclusive but suggests that such supplementation will decrease infant mortality from infectious disease through 6 m of age. The biological mechanism underlying this potential benefit is unclear but is presumed to include improving immune function. The investigators hypothesize that vitamin A supplementation at birth prevents vitamin A deficiency during a critical window of a few days to weeks when the immune system is first exposed to both normal, non-pathogenic organisms (e.g., commensal gut flora) and to potential pathogens. During this period the investigators propose that vitamin A supplementation will improve three aspects of immune function that will have sustained benefits throughout infancy: (1) normal thymus maturation and function; (2) development and mucosal targeting of adaptive immune responses, including regulatory T-cells (Treg), T-helper type 2 (Th2) cells, and IgA-secreting plasma cells and memory B-cells; and (3) mucosal barrier function. The three specific objectives of our project are: (1) Determine if vitamin A supplementation improves thymus maturation and function as indicated by ultrasonic analysis of thymus size and by analysis of thymic output of naïve T-cells using flow cytometric analysis of peripheral blood T-cells and by quantification of T-cell-receptor excision circles (TRECs) in peripheral blood. (2) Determine if vitamin A supplementation at birth alters (2.1) the T-cell response to BCG and OPV immunization assessed at 6 and 15 wk of age; (2.2) the T- and B-cell response to OPV immunization, assessed at 15 wk of age, and the secretory IgA response to OPV assessed at 6, 11 and 15 wk of age; and (2.3) the B-cell response to tetanus toxoid (TT) immunization, assessed at 15 wk of age. (3) Determine if vitamin A supplementation at birth will decrease bacterial lipopolysaccharide (LPS) concentrations in capillary blood, a marker of bacterial translocation.

ELIGIBILITY:
Inclusion Criteria:

* Infant receiving OPV and BCG within 48 hr of birth

Exclusion Criteria:

* Mother is less than 18 years of age
* Infant is part of a multiple birth
* Infant will likely not remain in the study area for the next 4 months
* Infant has a condition precluding vaccination
* Infant is unable to breastfeed or drink other fluids
* Birth weight is less than 1.5 kg

Max Age: 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Thymus size measured by ultrasound | through 15 wk of age
  Thymus size will be assessed sonographically using a validated method in which the transverse diameter of the thymus and the sagittal area of its largest lobe are multiplied to give a volume-related thymic index (TI). This index has been shown to correlate with thymus weight and has been used to show that the human thymus is sensitive to environmental influences during infancy.
peripheral blood naive T-helper lymphocyte concentration | through 15 wk of age
  Naive and memory CD4 T lymphocytes will be measured by flow cytometric analysis using the CD45RA and CD45RO markers to identify naive and memory CD4+ T-cells, respectively. Naive T cells develop in the thymus and their level in peripheral blood is an index of thymic function.
T-cell receptor excision circle (TREC) level in peripheral blood mononuclear cells (PBMC) | through 15 wk of age
  Thymic T-cell production can be assessed by measuring signal-joint T cell receptor excision circles (TRECs) as a traceable molecular marker in newly produced naive T-cells. Thus, the content of TRECs in peripheral blood is an indicator of thymopoiesis or newly synthesized and exported naive T-cells. TREC assessment will be conducted in the stored peripheral blood mononuclear cells (PBMC) isolated from infant's blood by standard Ficoll density gradient methods.
T-cell response to BCG (Bacillus Calmette-Guérin; to protect against tuberculosis) and oral polio virus (OPV) immunization | through 15 wk of age
  The Flow-cytometric Assay of Specific Cell-mediated Immune response in Activated whole blood (FASCIA) will be used on peripheral blood mononuclear cells to determine the percentage of CD4+ T cells that that are responsive to the BCG and OPV vaccines given at birth (OPV is given again at 6, 10 and 14 wk of age). The BCG response will be elicited using purified protein derivative of M. tuberculosis and the OPV response using formalin-inactivated polio virus antigen (types 1, 2 and 3).
Antibody response to oral polio virus (OPV) immunization | through 15 wk of age
  The antibody in lymphocyte supernatant (ALS) assay will be used to assess the production of polio-specific antibody by peripheral blood mononuclear cells (PBMC) at 15 wk of age and the secretory IgA response to OPV will be assessed at 6, 11 and 15 wk of age by measuring antibody in stool
T-cell and antibody response to tetanus toxoid (TT) and hepatitis B virus (HBV) vaccinations given at 6, 10 and 14 wk of age | through 15 wk of age
  The Flow-cytometric Assay of Specific Cell-mediated Immune response in Activated whole blood (FASCIA) will be used to measure the T-cell response to TT and HBV immunization using these vaccine antigens to stimulate a response at 6 and 15 wk of age. The antibody in lymphocyte supernatant assay (ALS) will be used to measure the antibody responses to these vaccines at 15 wk of age.
bacterial translocation to blood | through 15 wk of age
  Bacterial lipopolysaccharide (LPS) concentrations will be measured in plasma as a marker of bacterial translocation.

SECONDARY OUTCOMES:
vitamin A status by modified, relative dose-response (MRDR) test | through 15 wk of age
  vitamin A status will be measured using the MRDR in a subset of 30 subjects in each study arm.
bulging fontanelle | 48 h after vitamin A dosing
  The crainial fontanelle will be examined by study personnel to identify "bulging" as in indication of increased intracranial volume.

CONTACTS AND LOCATIONS:
Overall Officials: Charles B. Stephensen, Ph.D., Principal Investigator — USDA, Western Human Nutrition Research Center
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh

REFERENCES:
- [Derived] Ahmad SM, Huda MN, Raqib R, Qadri F, Alam MJ, Afsar MNA, Peerson JM, Tanumihardjo SA, Stephensen CB. High-Dose Neonatal Vitamin A Supplementation to Bangladeshi Infants Increases the Percentage of CCR9-Positive Treg Cells in Infants with Lower Birthweight in Early Infancy, and Decreases Plasma sCD14 Concentration and the Prevalence of Vitamin A Deficiency at Two Years of Age. J Nutr. 2020 Nov 19;150(11):3005-3012. doi: 10.1093/jn/nxaa260. PMID 32939553
- [Derived] Ahmad SM, Raqib R, Huda MN, Alam MJ, Monirujjaman M, Akhter T, Wagatsuma Y, Qadri F, Zerofsky MS, Stephensen CB. High-Dose Neonatal Vitamin A Supplementation Transiently Decreases Thymic Function in Early Infancy. J Nutr. 2020 Jan 1;150(1):176-183. doi: 10.1093/jn/nxz193. PMID 31504694
- [Derived] Huda MN, Ahmad SM, Alam MJ, Khanam A, Kalanetra KM, Taft DH, Raqib R, Underwood MA, Mills DA, Stephensen CB. Bifidobacterium Abundance in Early Infancy and Vaccine Response at 2 Years of Age. Pediatrics. 2019 Feb;143(2):e20181489. doi: 10.1542/peds.2018-1489. PMID 30674610
- [Derived] Ahmad SM, Raqib R, Qadri F, Stephensen CB. The effect of newborn vitamin A supplementation on infant immune functions: trial design, interventions, and baseline data. Contemp Clin Trials. 2014 Nov;39(2):269-79. doi: 10.1016/j.cct.2014.09.004. Epub 2014 Sep 28. PMID 25269669